CLINICAL TRIAL: NCT05380570
Title: Health Effects Associated With Occupational Radiation Exposure Among Korean Radiation Workers (Korean Radiation Workers Study)
Brief Title: Epidemiological Study of Korean Radiation Workers
Acronym: KRWS
Status: Active, not recruiting | Type: Observational
Sponsor: Korea Institute of Radiological & Medical Sciences (Other Government)
Responsible Party: Sponsor
Other Study IDs: 50091
Record Dates: First submitted 2022-05-09; First posted 2022-05-19 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Occupational Exposure to Radiation; Neoplasms, Radiation-Induced; Leukemia, Radiation-Induced; Radiation Effects
Keywords: Ionizing radiation; Cohort study; Radiation workers; Radiation-Induced diseases
MeSH Terms: conditions — Neoplasms, Radiation-Induced; Leukemia, Radiation-Induced

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Korean radiation workers: The study population is Korean radiation workers exposed to ionizing radiation in workplaces. Diagnostic medical radiation workers were not included in the study population.
  Interventions: Radiation: Occupational radiation exposure

INTERVENTIONS:
Radiation: Occupational radiation exposure — Ionizing radiation in workplaces

SUMMARY:
Health risks of radiation exposure in the moderate-to-high dose range have been well established. However, the risk remains unclear at low-dose ranges with protracted low-dose rate exposure, which is typical of occupational exposure. The purpose of this study is to construct a cohort of Korean radiation workers and to assess health effects associated with occupational radiation exposure. The study population is expected to be about 190,000 Korean radiation workers who have been registered with the Nuclear Safety and Security Commission since 1984. The national dose registry, the national cancer registry, the national vital statistics registry, and the national health insurance data are collected based on the Nuclear Safety Act. Through the linkage of those collected data, we will evaluate radiation-induced health risks including cancer and non-cancer diseases.

DETAILED DESCRIPTION:
The study population of this study is approximately 190000 Korean radiation workers registered with the Nuclear Safety and Security Commission since 1984. Diagnostic medical radiation workers were not included in the study population. The national dose registry, the national cancer registry, the national vital statistics registry, and the national health insurance data for radiation workers are collected retrospectively or prospectively based on the Nuclear Safety Act. Through the linkage of those collected data, we will evaluate radiation-induced health risks including cancer and non-cancer diseases. This data collection will be continued at 5-year intervals to update information on existing study participants and recruit newly hired workers if possible.

Age- and sex-specific standardized incidence and mortality ratios will be calculated for overall comparisons of cancer and non-cancer disease risks with general population. For dose-response assessment, excess relative risk (per Gy) and excess absolute risk (per Gy) will be estimated with adjustments for age and potential confounders, such as lifestyle factors and socioeconomic status.

ELIGIBILITY:
Inclusion Criteria:

* Korean radiation workers in the national dose registry (except for diagnostic medical radiation workers)

Exclusion Criteria:

* Unidentified personal identification numbers
* Foreigner

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Korean radiation workers in the national dose registry
Sampling Method: Non-Probability Sample
Enrollment: 196379 (Actual)
Dates: Start 2021-11-18 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2031-03-31 (Estimated)

PRIMARY OUTCOMES:
Radiation-induced cancer risk | year 4
  Cancer risk associated with occupational radiation exposure
Radiation-induced cancer risk | year 9
  Cancer risk associated with occupational radiation exposure

SECONDARY OUTCOMES:
Radiation-induced non-cancer risk | year 4
  Non-cancer disease risk associated with occupational radiation exposure
Radiation-induced non-cancer risk | year 9
  Non-cancer disease risk associated with occupational radiation exposure

CONTACTS AND LOCATIONS:
Locations (1):
- Korea Institute of Radiological & Medical Sciences, Seoul, Nowon-gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Seo S, Lim WY, Lee DN, Kim JU, Cha ES, Bang YJ, Lee WJ, Park S, Jin YW. Assessing the health effects associated with occupational radiation exposure in Korean radiation workers: protocol for a prospective cohort study. BMJ Open. 2018 Mar 30;8(3):e017359. doi: 10.1136/bmjopen-2017-017359. PMID 29602835
- [Result] Lee D, Cha ES, Park S, Sung H, Noh E, Jeong H, Jang WI, Seo S. Cohort Profile: The Korean Radiation Workers Study (KRWS). Int J Epidemiol. 2024 Apr 11;53(3):dyae060. doi: 10.1093/ije/dyae060. No abstract available. PMID 38628072